CLINICAL TRIAL: NCT01655979
Title: Medium-term Bedrest Whey Protein (MEP)
Acronym: MEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Collaborators: European Space Agency (Other); University Hospital, Clermont-Ferrand (Other); Institut Pluridisciplinaire Hubert Curien, Strasbourg, France (Unknown); Charite University, Berlin, Germany (Other); University of Milan (Other); Université de Nice Sophia Antipolis (Other); University of Ottawa (Other); Manchester Metropolitan University (Other); University of Toronto (Other); Medical University of Graz (Other); University of Cologne (Other); Radboud University Medical Center (Other); University Hospital, Lille (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ESA-AO-06-BR
Record Dates: First submitted 2012-07-23; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Countermeasure Evaluation
MeSH Terms: interventions — Whey Proteins; potassium bicarbonate

ARMS (2):
- MEP-1 (Experimental)
  Interventions: Dietary Supplement: Whey Protein + Potassium bicarbonate; Other: Control
- MEP-2 (Experimental)
  Interventions: Dietary Supplement: Whey Protein + Potassium bicarbonate; Other: Control

INTERVENTIONS:
Dietary Supplement: Whey Protein + Potassium bicarbonate — 0.6 mmol WP/kg body weight + 90 mmol KHCO3 during bed rest
Other: Control — Bed rest without dietary supplement

SUMMARY:
The human being has shown that he can live and work in the space environment, but due to the lack of essential mechanical load on muscle and bone, the fluid-shift as well as alterations in the acid-base balance (mainly on account of nutritional factors), the exposure to microgravity results in a gradual degradation of muscle, bone and cartilage, deconditioning of the cardiovascular system and metabolic changes. Countermeasures to prevent all the deconditioning of the physiological systems are not yet fully effective and require further investigation.

A commonly utilized model of simulating the physiological effects of microgravity on the human organism on ground is the 6° head-down-tilt bed rest. In the present study the model has been used to study potential countermeasures to spaceflight-associated deconditioning.

One of the most constrictive changes appearing during space flight as well as during bed rest, are disuse-induced muscle losses. These are associated with a decrease in muscle protein synthesis, rather then an increase in muscle protein breakdown. Besides an effective training countermeasure, nutritional countermeasures gain respect in this context: supplementing conventional diets with whey protein or essential amino acids has been shown to increase muscle protein synthesis. Due to these anabolic properties whey protein seems promising to counteract disuse-induced muscle wasting.

Drawbacks of a high protein intake are calciuric effects, ascribed to the proton-release when metabolizing sulfur-containing amino acids. The so called 'low grade metabolic acidosis' has also shown to activate osteoclastic bone resorption and muscle protein degradation. Therefore, to maximize the anabolic potential of a whey protein supplementation, the acidogenic properties need to be compensated. As previous works suggest, a shift of acid base balance into the acid direction and the resulting changes in bone and protein turnover may be hindered by supplementing alkaline mineral salts.

In this regard, a mid-term bed rest study was performed in order to investigate the effect of a combined whey protein (0.6 g/kg body weight/day) and potassium bicarbonate (90 mmol/day) supplementation as a potential countermeasure to multiple physiological and metabolic alterations on the human body resulting from real and simulated microgravity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, 20 -45 years
* BMI: 20 - 25 kg/m2
* Height: 158 - 190 cm
* Weight: 65 - 85 kg
* maximum relative oxygen uptake: 30 - 60 ml/min/kg
* non-smokers
* successful medical and psychological screening
* Willingness to participate in the entire study
* signed informed consent
* social insurance
* Clear criminal background check

Exclusion Criteria:

* Abuse of drugs, medicine or alcohol
* Vegetarians, Vegans
* Migraines
* History of mental illness
* Claustrophobia
* History of: thyroid dysfunction, renal stones, diabetes, allergies, hypertension, hypocalcaemia, uric acidaemia, lipidaemia, hyperhomocysteinaemia
* Rheumatism
* Muscle-, Cartilage- or Joint Injuries
* Gastro-esophageal reflux disease, renal function disorder, Hiatus hernia
* Chronic back pain
* Bone diseases
* Herniated discs
* Achilles tendon injuries
* Cruciate ligament rupture or any other severe knee injury
* BMD more than 1.5 SD < t-score
* History of orthostatic intolerance or vestibular disorders
* Anaemia
* Vitamin D Deficiency
* Positive response in thrombosis screening
* Use of metallic implants, osteosynthesis material
* Porphyria, Blood dyscrasia
* HIV, Hepatitis
* Increased Inner Eye pressure
* Intolerance to local anesthetics
* Participation in another study up to three month before study onset

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in body composition | Baseline, after 21 days of bed rest

SECONDARY OUTCOMES:
Plasma Volume | Baseline, after 21 days of bed rest
Maximum volume of oxygen uptake | Baseline, after 21 days of bed rest
Isometric torque | Baseline, after 21 days of bed rest
  During a an Isometric Maximum Voluntary Contraction Test on the knee extensors & flexors, the plantarflexors and dorsiflexors, the elbow extensors & flexors the Isometric Torque will be measured in Nm.
Muscle fatigue | Baseline, after 21 days of bed rest
Bone metabolism | Baseline, after 2,5,14,21 days of bed rest, 1, 5, 14, 28 days after finishing bed rest
Bone mineral density + content | Baseline, after 21 days of bed rest
Standing balance | Baseline, after 21 days of bed rest
Locomotion | Baseline, after 21 days of bed rest
  Locomotion will be assessed by Dynamic Gait Index, specific parameters are: total Score and Subscore
Body mass | Daily for a duration of 35 days
Intracranial pressure | Baseline, after 1,4, 7,10,13,14,15,16,17,18,19,20,21 days of bed rest,1,2,4 days after finishing bed rest
Monitoring of Vitamin K status | Baseline, after 2,5,14,21 days of bed rest, 1, 5 days after finishing bed rest
Fat metabolism | Baseline, after 21 days of bed rest
Glucose metabolism | Baseline, after 21 days of bed rest, 4 days after finishing bed rest
Nitrogen balance | Daily for a duration of 33 days
Energy metabolism | Baseline, after 21 days of bed rest
Glucocorticoid activity | Baseline, after 2,3,7,8,12,13,16,17 days of bed rest, 2,3 days after finishing bed rest
Muscle metabolism | Baseline, after 21 days of bed rest
Acid base balance | Baseline, after 2, 14, 21 days of bed rest, 5 days after finishing bed rest
Sympathetic activity during orthostatic stress | Baseline, after 21 days of bed rest
  Muscle sympathetic nerve activity is measured by MSNA recording by microneurography technique.
Visual Orientation | Baseline, after 6,12,20 days of bed rest, 2,4 days after finishing bed rest
  Visual Orientation is assessed by 'Oriented Character Recognition Test' and Luminous Line Test. The main parameter is Score.
Plasma galanin and adrenomedullin responses during head up tilt test (orthostatic stress) | Baseline, after 21 days of bed rest
Cartilage metabolism and -thickness | Baseline, after 2,3,5,7,14,21 days of bed rest, 5 days after finishing bed rest
Hematopoetic system | Baseline, after 10, 21 days of bed rest, 1, 28 days after finishing bed rest
  Blood cell count, reticulocytes, Haptoglobin, Bilirubin, Ferritin, EPO, Thrombopoietin, Urinary Urobilinogen and Fecal Urobilinogen (markers of blood cell degradation)
Fat accumulation in bone marrow | Baseline, after 10, 21 days of bed rest, 3, 28 days after finishing bed rest
Achilles tendon structure | Baseline, after 21 days of bed rest, 2, 28 days after finishing bed rest
Headache - frequency and quality | Baseline, daily during 21 days of bed rest
Muscle volume | Baseline, after 20, 21 days of bed rest, 3 days after finishing bed rest
Free water and fat content in muscle | Baseline, after 20, 21 days of bed rest, 3 days after finishing bed rest
Orthostatic tolerance | Baseline, after 21 days of bed rest
  Orthostatic tolerance will be assessed by Head up tilt test. The following parameters are assessed to measure orthostatic tolerance: beat-to-beat heart rate [bpm], beat-to-beat blood pressure [bpm] time to presyncope [min, s]

CONTACTS AND LOCATIONS:
Locations (1):
- DLR German Aerospace Center, Cologne, Germany

REFERENCES:
- [Derived] Rudwill F, O'Gorman D, Lefai E, Chery I, Zahariev A, Normand S, Pagano AF, Chopard A, Damiot A, Laurens C, Hodson L, Canet-Soulas E, Heer M, Meuthen PF, Buehlmeier J, Baecker N, Meiller L, Gauquelin-Koch G, Blanc S, Simon C, Bergouignan A. Metabolic Inflexibility Is an Early Marker of Bed-Rest-Induced Glucose Intolerance Even When Fat Mass Is Stable. J Clin Endocrinol Metab. 2018 May 1;103(5):1910-1920. doi: 10.1210/jc.2017-02267. PMID 29546280